CLINICAL TRIAL: NCT05947617
Title: Phase 1 Study: Assessing VIX001 Safety, Efficacy, and Dosing in Post Acute COVID-19 Syndrome (PACS) Patients With Neurological Symptoms and Cognitive Impairment.
Brief Title: Safety, Efficacy, and Dosing of VIX001 in Patients With Neurological Symptoms of Post Acute COVID-19 Syndrome (PACS).
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neobiosis, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IND_28592; VIX001-PACS-01 (Other: Neobiosis,LLC)
Record Dates: First submitted 2023-07-11; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Post-Acute COVID-19 Syndrome; Cognitive Impairment; Neurological Complication
Keywords: Post-Acute COVID-19 Syndrome (PACS); Cognitive Impairment; Amniotic Fluid Product; VIX001; Neurological Symptoms; Phase 1 Trial; Dose-Escalation Study; Safety; Tolerability; Preliminary Efficacy; Dose Effect; Intravenous Injection; SARS-CoV-2 Infection; Montreal Cognitive Assessment (MoCA)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cognitive Dysfunction; Neurologic Manifestations; COVID-19

STUDY DESIGN:
Intervention Model Description: The study follows a dose-escalation design where participants are enrolled in sequential cohorts receiving escalating doses of VIX001 (1 ml, 3 ml, or 10 ml). This suggests a sequential approach in terms of dose administration within the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Low Dose (1 ml) VIX001 (Experimental): Participants in this arm will receive intravenous injections of VIX001 at a low dose of 1 ml. The intervention involves the administration of VIX001 diluted in clinical standard saline.
  Interventions: Drug: VIX001
- Arm 2: Intermediate Dose (3 ml) VIX001 (Experimental): Participants in this arm will receive intravenous injections of VIX001 at an intermediate dose of 3 ml. The intervention entails the administration of VIX001 diluted in clinical standard saline.
  Interventions: Drug: VIX001
- Arm 3: High Dose (10 ml) VIX001 (Experimental): Participants in this arm will receive intravenous injections of VIX001 at a high dose of 10 ml. The intervention involves the administration of VIX001 diluted in clinical standard saline.
  Interventions: Drug: VIX001

INTERVENTIONS:
Drug: VIX001 — This study utilizes a dose-escalation design with three arms or cohorts to evaluate the safety, tolerability, preliminary efficacy, and dose effect of VIX001, an amniotic fluid product, in patients with Post-Acute COVID-19 Syndrome (PACS) associated with neurological symptoms of cognitive impairment.
  In all arms, the intervention will be administered at baseline and participants will be assessed at specified timepoints for safety, cognitive impairment, pain, activity, and quality of life. The primary objective is to evaluate the safety of VIX001, while the secondary objectives include assessing its potential efficacy and patient-reported outcomes.
  Other Names: Purified Amniotic Fluid

SUMMARY:
The study, identified as VIX001-PACS-01, is a Phase 1, open-label, dose-escalation trial evaluating the safety, tolerability, preliminary efficacy, and dose effect of VIX001, an amniotic fluid product, in patients with Post-Acute COVID-19 Syndrome (PACS) and cognitive impairment. Conducted at the University of Miami Hospital and Clinics, the trial aims to enroll up to nine participants, or up to 18 using a 3+3 dose escalation design. Intravenous injections of VIX001 will be administered at three ascending doses (1 ml, 3 ml, or 10 ml), and participants will be assessed for safety, cognitive impairment, pain, activity, and quality of life at baseline and various timepoints. The primary objective is to evaluate the safety of VIX001, while secondary objectives include assessing its potential efficacy and patient-reported outcomes. The study duration is expected to last approximately 18 months, including enrollment, evaluation, and post-study observation periods. The findings will contribute to understanding VIX001's safety and efficacy in treating PACS-related cognitive impairment.

DETAILED DESCRIPTION:
Study Title: A Phase 1, Open-label Dose-Escalation Study to Assess the Safety, Tolerability, Preliminary Efficacy, and Dose Effect of VIX001 Amniotic Fluid Product in Patients with Post-Acute COVID-19 Syndrome (PACS) Associated with Neurological Symptoms of Cognitive Impairment

Study Number: VIX001-PACS-01

Study Design: This is a Phase 1, open-label, dose-escalation trial aimed at evaluating the safety, tolerability, preliminary efficacy, and dose effect of VIX001, an amniotic fluid product, in patients with Post-Acute COVID-19 Syndrome (PACS) who are experiencing neurological symptoms of cognitive impairment. The study will follow a 3+3 dose escalation design, with up to nine participants enrolled initially, and a possibility of expanding to up to 18 participants if toxicities occur within the predefined dosing range.

Study Objectives: The primary objective of the study is to assess the safety of VIX001 when administered intravenously to patients with PACS and cognitive impairment. The secondary objectives include evaluating the preliminary efficacy of VIX001 on cognitive impairment, pain, activity, and quality of life in these patients.

Study Center: The study will be conducted at the University of Miami Hospital and Clinics.

Study Duration: The anticipated duration of the study is approximately 18 months. This includes a six-month enrollment period, a six-month evaluation period for each participant, and a six-month post-study observation period.

Participant Eligibility Criteria: To be eligible for the study, participants must have a prior laboratory-confirmed SARS-CoV-2 infection, a recent negative SARS-CoV-2 test, and have experienced moderate or severe post-COVID-19 symptoms for a minimum of three months. Participants should exhibit reduced physical functioning compared to their pre-COVID-19 status and present with neurological impairment, as indicated by a score of ≤ 24 on the Montreal Cognitive Assessment (MoCA).

Investigational Product: VIX001 is an amniotic fluid product derived from qualified donors. It will be administered intravenously at three ascending doses: 1 ml, 3 ml, or 10 ml. VIX001 will be diluted in clinical standard saline for administration.

Study Procedures: Participants will receive intravenous injections of VIX001 at the assigned dose level. Safety evaluations, including medical history, physical examinations, and selected laboratory tests, will be conducted at specified timepoints. Cognitive impairment, pain, activity, and quality of life will also be assessed using validated measures at baseline and at multiple timepoints during the study.

Endpoints: The primary endpoint of the study is the safety of VIX001, which will be evaluated by monitoring treatment-emergent adverse events. The secondary endpoints include changes in cognitive impairment and various patient-reported outcomes related to PACS, such as pain, activity levels, and quality of life.

Planned Participant Number: The study aims to enroll up to nine participants initially, or up to 18 participants if toxicities occur within the predefined dosing range.

This Phase 1 clinical trial aims to assess the safety, tolerability, preliminary efficacy, and dose effect of VIX001, an amniotic fluid product, in patients with PACS and cognitive impairment. The findings will contribute to understanding the potential of VIX001 as a therapeutic intervention for patients with neurological symptoms associated with PACS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Has had prior laboratory-confirmed SARS-CoV-2 infection as determined by an approved polymerase chain reaction (PCR) or an approved antigen test of any specimen, which did not require intubation or mechanical or non-invasive ventilation to address the SARS-CoV-2 infection. Only those who had COVID-19 and who were not hospitalized for their infection and are eligible for this study.
3. Has had a recent (within a week) negative SARS-CoV-2 test (an approved PCR or antigen test).
4. Has had at least moderate or severe post-COVID-19 symptoms for at least 3 months which have resulted in reduced functioning compared to pre-COVID-19 status, and a working diagnosis of post-acute COVID-19 syndrome (PACS).
5. Ability to comply with the requirements of the study, including anticipated ability to attend all scheduled visits.
6. Ability to understand and provide written informed consent.
7. All participants of reproductive age/capacity will be required to use adequate contraception, defined as two forms of highly effective contraceptives, with any partners during the study period and for at least three months beyond the study period for safety.
8. The primary presenting symptom impeding daily function is neurological.
9. Severity of cognitive impairment/brain fog measured by MoCA score of ≤ 24 [40] that was not present prior to contracting COVID-19. A score of 18-26 indicates mild cognitive impairment. A score of 17 or less may indicate moderate impairment. This study will enroll patients with so-called "brain fog," or mild impairment to the degree that would not affect capacity to consent. A careful history will be taken to ensure that the symptoms of cognitive impairment found to be limiting by the patient and their family (if applicable) have developed subsequent to the COVID-19 infection, and were not present previously. If the temporal course of the clinical history is not clearly related to the acute infection, the patient will not be considered for inclusion. In parallel, the following neurological symptoms will be assessed and monitored as exploratory endpoints, but are not inclusion criteria:

   * Objective assessment of orthostatic intolerance as determined by a change of 30 in pulse or blood pressure on NASA 10-Minute Lean Test in patients who had no prior history of autonomic dysfunction;
   * Symptomatic depression (defined as a score of <10 on the PHQ-8 patient reported outcome questionnaire) at the time of screening that must have been controlled on a stable therapy (pharmacological or in the care of a therapist) for three months prior to planned infusion, are under the active care of a mental health provider during the study period, and was not present prior to contracting COVID-19.;
   * Anxiety on GAD-7 with a score of ≥10 and ≤ 15 that was not present prior to contracting COVID-19; and
   * Sleep disturbance on PROMIS-SD with a score of ≥30 that was not present prior to contracting COVID-19.

Exclusion Criteria:

1. Significant concurrent medical conditions (verified by medical records as needed), including the following:

   * Poorly controlled diabetes mellitus, defined as HbA1C>8.5.
   * Medical History of Chronic kidney disease (CKD) diagnosis and/or screening results of eGFR < 60mL/min/1.73m2.
   * Presence of New York Heart Association (NYHA) Class III/IV heart failure during screening visit.
   * Blood pressure > 180/110 mm/Hg during screening visit.
   * Chronic obstructive pulmonary disease (COPD).
   * Participants with HIV, Hepatitis B and Hepatitis C.
2. Participants with a prior history of stroke, neurogenerative disease, dementia, or developmental delay.
3. Participants with < 18 on MoCA will be excluded, as well as any who have an active power of attorney or other legal basis to be deemed to lack capacity.
4. Participants who require ongoing oxygen ventilation.
5. Other clinically significant, ongoing illness or medical condition, that in the opinion of the investigator constitutes a safety risk for participation in the study or that could interfere with achieving the study objectives, conduct or evaluation, including a history of thromboembolic events.
6. Participants who are pregnant or lactating.
7. Active alcohol or substance abuse or any other reason that makes it unlikely that the participant will comply with study procedures.
8. Infusion of any other investigational agents within 6 months of randomization.
9. All subjects with PHQ-8 score >10 at the time of enrollment screening will be excluded from the study.
10. Participants with a psychiatric illness or condition, which, in the opinion of the investigation, would interfere with the conduct of the study or the interpretation of study results. Participants with stable anxiety and depression (PHQ-8 score of <10) defined as being on stable doses of antidepressant and anxiety drugs for the last 3 months and for which no dose changes are expected during the study can be included. Participants who are not under the active care of a mental health provider during the study period will be excluded.
11. Participants with autoimmune disease or a known history of having Acquired Immunodeficiency Syndromes (AIDS) or Human Immunodeficiency Virus (HIV).
12. Participant has known alcoholic addiction or dependency, uses alcohol daily, or has current substance use or abuse.
13. Participant has any active malignancy, including evidence of cutaneous basal, squamous cell carcinoma, or melanoma.
14. Participant was either diagnosed with or reasonably believed to have had Chronic Fatigue Syndrome, Sleep Apnea, Insomnia, or any other sleep disorder prior to contracting COVID-19.
15. Significant laboratory abnormalities, including any of the following

    * White blood cell count < 3000/mm3.
    * Platelet count < 125,000 mm3.
    * Absolute neutrophil count < 1500/mm3.
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN) x 1.5.
    * any other laboratory abnormality, which, in the opinion of the investigator poses a safety risk or will prevent the participant for completing the study.
    * Uncontrolled Hyperthyroidism or Hypothyroidism or any other Thyroid disease reflected by abnormal TSH per local laboratory. Those with abnormal TSH in conjunction with either an abnormal T3 or Free T4 will be excluded.
16. Recent vaccination against SARS-CoV-2 within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Six Minute Walk Test (6MWT) with oximetry. | Day 0, 7, 30, 90, 180
  Physiologic assessments
Change from Baseline Transthoracic Echocardiogram in 3 Dimensions (3-D TTE). | Day 30, 90, 180
  Physiologic assessments
Change from Baseline Pulmonary Function Test (PFT) with bronchodilation if abnormal. | Day 30, 90, 180
  Physiologic assessments
Change from Baseline Sleep time and depth parameters derived from wearable device (Biostrap). | Day 180
  Physiologic assessments
Change from Baseline Heart Rate Variability (HRV) during sleep, derived from wearable device (Biostrap). | Day 180
  Physiologic assessments
Change from Baseline UPSIT testers. | Day 30, 90, 180
  Physiologic assessments
Change from Baseline Montreal Cognitive Assessment (MoCA). | Day 0, 7, 30, 90, 180
  Physiologic assessments
Change from Baseline NASA 10-Minute Lean Test. | Day 7, 30, 90, 180
  Physiologic assessments
Change from Baseline CNS Vital Signs test battery. | Day 7, 30, 90, 180
  Physiologic assessments

SECONDARY OUTCOMES:
PROMIS | Day 0, 7, 30, 90, 180
  Patient-Reported outcomes
  1. Sleep Disturbance
  2. Fatigue
  3. Physical Function
  4. Pain Interference
mMRC Scale. | Day 0, 7, 30, 90, 180
  Patient-Reported outcomes
General Anxiety Disorder (GAD-7). | Day 0, 7, 30, 90, 180
  Patient-Reported outcomes
Personal Health Questionnaire Depression Scale (PHQ-8). | Day 0, 7, 30, 90, 180
  Patient-Reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Roger Alvarez, DO, MPH, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No
The principal investigator must maintain all documentation related to the study for a period of two years after the last marketing application approval, or if not approved, two years following the discontinuance of the test article for investigation. If it becomes necessary for the sponsor or the regulatory authority to review any documentation related to the study, the investigator must permit access to such records.